CLINICAL TRIAL: NCT00888940
Title: CONSERV - 2 (Clinical Outcomes and Safety Trial to Investigate Ecallantide's Effect on Reducing Surgical Blood Loss Volume) - A Phase 2 Randomized Double-Blind Active-Controlled Study in Subjects Exposed to Cardio-pulmonary Bypass During Cardiac Surgery at High Risk of Bleeding
Brief Title: Outcomes and Safety Trial Investigating Ecallantide's Effect on Reducing Surgical Blood Loss Volume in Subjects at High Risk of Bleeding Exposed to Cardio-pulmonary Bypass During Cardiac Surgery
Acronym: CONSERV-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECAL-CCPB-08-07
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Results first posted 2011-01-17 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Bloodloss; Surgical Procedures, Operative
MeSH Terms: interventions — ecallantide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ecallantide (Experimental)
  Interventions: Drug: Ecallantide
- Cyklokapron(R) (Active Comparator)
  Interventions: Drug: Cyklokapron(R)

INTERVENTIONS:
Drug: Ecallantide — 2.25 mg/L pump prime, 0.13 mg/kg loading dose, 2.25 mg/L constant infusion
  Arms: ecallantide
Drug: Cyklokapron(R) — 1000-mg loading dose followed by a continuous infusion of 400 mg/hr with an additional 500 mg added to the pump prime
  Arms: Cyklokapron(R)

SUMMARY:
A Phase 2 Randomized Double-Blind Active-Controlled Study in Subjects Exposed to Cardio-pulmonary Bypass During Cardiac Surgery at High Risk of Bleeding

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (by study subject) prior to any study-related procedure not part of normal medical care;
* Male or female between the ages of 18 and 85 years old, inclusive; and
* Planned cardiac surgery using cardio-pulmonary bypass, for one of the following procedures: any repeat sternotomy; surgery to repair or replace more than one valve; combined CABG plus repair or replacement of at least one valve
* If female, subject is non-lactating, and is either:Not of childbearing potential, defined as postmenopausal for at least one year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy, or hysterectomy;Of childbearing potential but is not pregnant as confirmed by negative pregnancy test at time of screening (based on the β-subunit of HCG), and is practicing the barrier method of birth control along with one of the following methods: oral or parenteral contraceptives for three months prior to study drug administration, a vasectomized partner, or abstinence from sexual intercourse.

Exclusion Criteria:

* Planned primary CABG, single valve repair or replacement surgery, or any off pump procedure;
* Body weight <55 kg;
* Planned hypothermia (<28ºC);
* Planned transfusion in the peri-operative or post-operative periods;
* Planned transfusion of pre-operatively donated autologous blood;
* Female subjects who are pregnant or lactating;
* Planned use of desmopressin, lysine analogs (other than study medication), atrial natriuretic hormone or recombinant activated Factor VII;
* Planned use of corticosteroids in the pump prime solution;
* Ejection fraction <30% within 90 days prior to surgery;
* Evidence of a myocardial infarction within 5 days prior to surgery;
* History of stroke or transient ischemic attack within 3 months prior to surgery;
* Hypotension or heart failure requiring the use of inotropes or mechanical devices within 24 hours prior to surgery;
* Serum creatinine >2.0 mg/dL within 48 hours prior to surgery;
* Serum hepatic enzymes (aspartate aminotransferase or alanine aminotransferase) above 2.5 times the upper limit of normal for the applicable laboratory;
* Hematocrit <32% within 48 hours prior to surgery;
* Platelet count below the normal range for the applicable laboratory within 14 days prior to surgery;
* History of, or family history of, bleeding or clotting disorder (e.g. von Willebrand's Disease, idiopathic thrombocytopenia purpura) or thrombophilia such as anti-thrombin III deficiency or Factor V Leiden mutation;
* History of heparin-induced thrombocytopenia;
* Prothrombin time (PT) and/or activated partial thromboplastin time (aPTT) >1.5 X normal range unless subject received heparin within 24 hours of test;
* Serious intercurrent illness or active infection (e.g. endocarditis, sepsis, active malignancy requiring treatment);
* Any previous exposure to ecallantide;
* Receipt of an investigational drug or device 30 days prior to participation in the current study;
* Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or would preclude the subject from successful completion of the study;
* Inability to comply with the protocol for the duration of the study;
* Known allergy to any agent expected to be used in the intra-operative or post-operative periods; and
* Administration of: Eptifibatide within 6 hours prior to surgery, Tirofiban hydrochloride within 6 hours prior to surgery, (Enoxaparin sodium or other low-molecular-weight heparin <24 hours prior to surgery), Prasugrel within 10 days prior to surgery, Clopidogrel within 3 days prior to surgery, Ticlopidine within 7 days prior to surgery, Abciximab within 5 days prior to surgery, (Bivalirudin, argatroban or lepirudin within 6 hours prior to surgery), (Fondaparinux within 72 hours prior to surgery), Chlorpromazine within 7 days prior to surgery (Prophylactic use permitted for the prevention of deep vein thrombosis.)
* Planned use of heparin bonded bypass circuits;
* Known allergy or hypersensitivity to tranexamic acid or any of the other ingredients;
* Disturbance of color sense;
* Evidence of hematuria or any acute thromboses or thromboembolic diseases such as deep vein thrombosis, pulmonary embolism, or vertebral vein thrombosis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alistair Wheeler, MD, MFPM, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (34):
- Cardio-Thoracic Surgeons PC, Birmingham, Alabama, United States
- Germany (20):
  - Universitaetsklinikum Aachen AoeR, Aachen
  - Klinikum Augsburg, Augsburg
  - Herz- und Gefaesszentrum Bad Bevensen, Bad Bevensen
  - Universitaetsklinikum Bonn, Bonn
  - Klinik und Poliklinik fuer Herz- und Thoraxchirurgie der Universitaet zu Koeln, Cologne
  - St. Johannes Hospital, Dortmund
  - Herzzentrum Dresden GmbH Universitaetsklinik, Dresden
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsmedizin Goettingen, Göttingen
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaeres Herzzentrum Hamburg GmbH, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Stadt Ludwigshafen gGmbH, Ludwigshafen
  - Klinik fuer Herzchirurgie des Universitaetsklinikum SH, Lübeck
  - Deutsches Herzzentrum Muenchen, Munich
  - HELIOS Klinik Wuppertal, Wuppertal
  - Universitaetsklinikum Wuerzburg, Würzburg
- Poland (13):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki im. Dr. Antoniego Jurasza w Bydgoszczy, Bydgoszcz
  - Akademickie Centrum Kliniczne, Szpital AM w Gdansku, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny nr 7 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Uniwersytecki Szpital Kliniczny Nr. 3 im. Dr Seweryna Sterlinga, Lódz
  - Katedra Chorób Serca AM, Szpital Miejski im. J Strusia, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 Pomorskiej Akademii Medycznej, Szczecin
  - Wojskowy Instytut Medyczny, Centralny Szpital Kliniczny MON, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiclecia Stefana Kardynała Wyszyńskiego, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Centrum Chorób Serca, Wroclaw
  - Slaskie Centrum Chorób Serca, Zabrze

REFERENCES:
- [Derived] Bokesch PM, Szabo G, Wojdyga R, Grocott HP, Smith PK, Mazer CD, Vetticaden S, Wheeler A, Levy JH. A phase 2 prospective, randomized, double-blind trial comparing the effects of tranexamic acid with ecallantide on blood loss from high-risk cardiac surgery with cardiopulmonary bypass (CONSERV-2 Trial). J Thorac Cardiovasc Surg. 2012 May;143(5):1022-9. doi: 10.1016/j.jtcvs.2011.06.001. Epub 2011 Jul 2. PMID 21724197

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ecallantide | Cyklokapron(R)
Started | 120 | 122
Completed Therapy | 107 | 106
Completed | 92 | 101
Not Completed | 28 | 21
Not completed — Adverse Event | 12 | 3
Not completed — Lost to Follow-up | 5 | 5
Not completed — Randomized Not Treated | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ecallantide | Cyklokapron(R) | Total
Number analyzed (Participants) | 120 | 122 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.02) | 66.9 (10.88) | 68.2 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 50 | 95
  Male | 75 | 72 | 147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 120 | 122 | 242
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Volume of Packed Red Blood Cells Transfused
Time Frame: 12 hours after the end of surgery
Population: Modified Intent to Treat = all subjects received at least one dose and analyzed according to planned treatment assignment. 3 subjects in ecallantide group not included due to no value being present
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ecallantide | Cyklokapron(R)
Number analyzed (Participants) | 106 | 109
mL | 1223.2 (1334.57) | 623.5 (974.64)
Statistical Analysis 1: Comparison: Ecallantide vs Cyklokapron(R); Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Treatment-emergent Adverse Events.
Time Frame: Over the duration of the study.
Population: Safety population analyzed
Measure: Number; unit: events
Arm/Group | Ecallantide | Cyklokapron(R)
Number analyzed (Participants) | 109 | 109
events
  At Least 1 TEAE | 100 | 94
  At Least 1 Related TEAE | 5 | 5
  At Least 1 Severe TEAE | 38 | 17
  At Least 1 Serious TEAE | 45 | 28
  At Least 1 Related & Serious TEAE | 4 | 1
  Premature Study Drug Discontinuations Due to TEAE | 2 | 2
  Related TEAE Resulting in Discontinuation of Drug | 0 | 0
  TEAE Resulting in Death | 13 | 4
  Related TEAE Resulting in Death | 0 | 0

ADVERSE EVENTS:
Groups:
- Cyklokapron: 1000-mg loading dose followed by a continuous infusion of 400 mg/hr with an additional 500 mg added to the pump prime
Arm/Group | Ecallantide | Cyklokapron
Serious Adverse Events (participants affected / at risk) | 45/109 | 28/109
Other Adverse Events (participants affected / at risk) | 93/109 | 91/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecallantide (N=109) | Cyklokapron (N=109)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 4 (4) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Ventricle rupture (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 1 (1)
Multi-organ failure (General disorders) | 3 (3) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 11 (13) | 7 (7)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac output decreased (Investigations) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0)
Impaired self-care (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 9 (9) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ecallantide (N=109) | Cyklokapron (N=109)
Anaemia (Blood and lymphatic system disorders) | 18 (18) | 16 (17)
Arrhythmia (Cardiac disorders) | 7 (7) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 32 (32) | 19 (20)
Tachycardia (Cardiac disorders) | 3 (3) | 9 (9)
Constipation (Gastrointestinal disorders) | 9 (9) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (8)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Vomiting (Gastrointestinal disorders) | 7 (8) | 4 (4)
Impaired healing (General disorders) | 6 (6) | 9 (9)
Non-cardiac chest pain (General disorders) | 7 (9) | 9 (10)
Oedema peripheral (General disorders) | 6 (6) | 7 (7)
Procedural pain (Injury, poisoning and procedural complications) | 17 (18) | 25 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (11) | 15 (15)
Sleep disorder (Psychiatric disorders) | 5 (5) | 6 (7)
Transient psychosis (Psychiatric disorders) | 7 (7) | 4 (4)
Renal failure (Renal and urinary disorders) | 3 (3) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 17 (17)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 6 (6) | 10 (10)
Hypotension (Vascular disorders) | 20 (20) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication is initiated by Cubist. If the First Publication is not published within 1 year of Study conclusion or termination, Investigator shall have the right to publish and disclose the Data. Prior to any submission for publication, presentation, or communication of results or information arising from the Study, Investigator shall provide Cubist at least 90 days for review and comment upon the manuscript or other material for such publication or presentation.